CLINICAL TRIAL: NCT07105631
Title: Patient-reported Outcomes (PRO) and Treatment Outcomes of Chinese Patients With MSS-type Advanced Colorectal Cancer Who Received the Zidovudine Combination Regimen in the Real World: A Prospective, Multicenter, Observational Study Protocol
Brief Title: Patient-reported Outcomes (PRO) and Treatment Outcomes of Chinese Patients With MSS-type Advanced Colorectal Cancer Who Received the Zidovudine Combination Regimen in the Real World
Status: Recruiting | Type: Observational
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, Meng Qiu, PhD, West China Hospital
Other Study IDs: CSIIT-Q108
Record Dates: First submitted 2025-05-20; First posted 2025-08-06 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-05

CONDITIONS: Colorectal Cancer
Keywords: HDAC inhibitors; pMMR/MSS; electronic patient-reported outcome; Real world study
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Chidamide+Immune checkpoint inhibitors+others: Chidamide+Immune checkpoint inhibitors+others

SUMMARY:
The Chidamide + sintilimab ± bevacizumab regimen has become a post-treatment option for clinicians and patients after being included in the guidelines. The CAPability-01 study is a phase II RCT, with a limited number of enrolled subjects. Further observation of the safety and clinical real-world application status of the sidibemab combination regimen is needed in a larger sample size prospective observational cohort study. The primary endpoint of this study is the safety events of the sidibemab combination regimen.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years old, gender not restricted;
2. Advanced colorectal cancer confirmed by histopathology; and confirmed as MSS/pMMR type by immunohistochemistry or genetic testing;
3. The investigators evaluate that the treatment regimen of cediranib combined with immune checkpoint inhibitors is applicable;
4. Clear consciousness, able to answer questions correctly;
5. Capable of using mobile phones and accessing the internet, with 3G/4G/5G function of smart mobile devices.

Exclusion Criteria:

1. There are serious complications that interfere with the efficacy and safety analysis;
2. The investigators determined that the subjects were not suitable for inclusion in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with MSS/pMMR advanced colorectal cancer treated with the Chidamide combined with ICI therapy regimen
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2025-07-10 (Actual); Primary Completion 2026-07-30 (Estimated); Study Completion 2027-07-30 (Estimated)

PRIMARY OUTCOMES:
Grade 3-4 adverse effects rate | From date of randomization until the date of death from any cause, assessed up to 2 years]
  Rate of HDACi and immunotherapy and others treatments related severe adverse events

SECONDARY OUTCOMES:
Objective response rate（ORR） | about a year
  Objective response is defined as a complete response (CR
  ) or partial response (PR) according to RECIST v.1.1 or iRECIST
Overall survival (OS) | 2 years
  Time from randomization to date of death due to any cause
  . according to the RECIST version 1.1 or iRecist recorded in the time period between randomization death to any cause.
Progression-free survival（PFS） | 2 years
  Time from randomization to date of Disease progression or death due to any cause.according to the RECIST version 1.1 or iRecist recorded in the time period between randomization and disease progression or death to any cause.
Duration of Response（DOR） | 2 years
  Time from randomization to date of the first assessment of the tumor as CR (Complete Response) or PR (Partial Response) until the first assessment of PD (Progressive Disease) or death for any reason.according to the RECIST version 1.1 or iRecist.
Clinical benefit rate （CBR） | 2 years
  Time from randomization to date of the first assessment of the tumor as CR (Complete Response) or PR (Partial Response) or SD (Stable Disease)rate.according to the RECIST version 1.1 or iRecist.

CONTACTS AND LOCATIONS:
Locations (1):
- West China Hospital Sichuan University, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No